CLINICAL TRIAL: NCT07104747
Title: A Comparative Study on The Effects of Static Versus Dynamic Exercises on Balance and Activity Balance Confidence In The Elderly Population With Locomotive Syndrome
Brief Title: The Effects of Static Versus Dynamic Exercises on Balance and Activity Balance Confidence In The Elderly Population With Locomotive Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Dr, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TUF/PB/33/1026/33
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Locomotive Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static Exercise Intervention (Experimental): Participants performed static balance exercises three times per week for six weeks, progressing in difficulty over time. In weeks 1-2, exercises were performed with support and included tandem standing, standing on a balance cushion, lunges with hand support, and one-leg stands. In weeks 3-4, the same exercises were done without support, and in weeks 5-6, they were performed with eyes closed to increase sensory challenge. Exercise duration progressed from 3 sets of 60 seconds to 5 sets of 90 seconds, and finally 7 sets of 120 seconds per movement.
  Interventions: Procedure: Static Exercise Intervention
- Dynamic Exercise Intervention (Active Comparator): This group engaged in dynamic balance exercises, also three times weekly for six weeks, with progressive complexity. Initial sessions (weeks 1-2) included walking with obstacles,tandem walking with support, small-step lunges, and supported step-ups.Weeks 3-4 incorporated cognitive elements and increased difficulty,while weeks 5-6 introduced sensory challenges like walking with eyes closed. Repetitions increased from 3sets of 60 seconds to 7 sets of 120 seconds, aligning with the progression in task complexity.
  Interventions: Procedure: (Dynamic Exercises Group

INTERVENTIONS:
Procedure: Static Exercise Intervention — Static exercises generally involve maintaining a fixed position without movement-such as standing on one leg or holding a specific posture-emphasizing isometric muscle control and stability.
  Arms: Static Exercise Intervention
Procedure: (Dynamic Exercises Group — Dynamic exercises were structured across three progressive stages-basic, moderate, and advanced-each increasing in complexity and difficulty. These exercises were performed in various positions, including sitting, standing, and walking.
  Arms: Dynamic Exercise Intervention

SUMMARY:
This research aimed to explore the comparative effects of static and dynamic balance training on postural stability and activity-specific balance confidence among elderly individuals diagnosed with locomotive syndrome. A single-blinded, randomized clinical trial was conducted at a shelter home, where thirty participants between the ages of 60 and 75 were randomly assigned to two intervention groups. One group received static balance exercises, while the other group engaged in dynamic balance training. Both interventions were delivered three times per week over a six-week period. Standardized assessment tools, including the Y-Balance Test and the Activities-specific Balance Confidence (ABC) Scale, were used to evaluate outcomes related to balance and self- perceived confidence in performing daily activities. The study was designed to determine the more effective approach for enhancing mobility and promoting independence in the elderly population affected by locomotive syndrome.

ELIGIBILITY:
Inclusion Criteria:

Able to walk independently People with locomotive syndrome Can be able to perform exercise and listen to the therapist

Exclusion Criteria:

* Any mental illness Any systemic Illness

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Y balance test | 6 weeks
  Y Balance Test larger reach distances and higher symmetry between limbs reflect greater dynamic balance and functional capacity

SECONDARY OUTCOMES:
Activity balance confidence | 6 weeks
  Activity-Specific Balance Confidence (ABC) Scale higher scores suggest an enhancement in patient confidence regarding balance in a range of daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Izza Ayub; PT, Faisalābad, Pakistan

IPD SHARING:
Plan to Share IPD: No